CLINICAL TRIAL: NCT03184818
Title: Outcomes of Urinary Tract Infection Management by Pharmacists
Acronym: RxOUTMAP
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Horizon Health Network (Other); New Brunswick Pharmacists' Association (Unknown); Loblaw Companies Ltd. (Unknown); Pharmasave Drugs (Atlantic) Ltd. (Unknown); Alberta Pharmacists Association (Unknown); The Jean Coutu Group (PJC) Inc. (Unknown)
Responsible Party: Principal Investigator, Ross T. Tsuyuki, Professor of Medicine (Cardiology) and Director, EPICORE Centre, University of Alberta, University of Alberta
Other Study IDs: Pro00072493
Record Dates: First submitted 2017-06-07; First posted 2017-06-14 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No antibacterial from other provider (Arm 1): Patients with symptomatic, uncomplicated urinary tract infection presenting without a prescription for an antibacterial from another health care practitioner.
  Interventions: Other: Advanced care
- Antibacterial from other provider (Arm 2): Patients with symptomatic, uncomplicated urinary tract infection or asymptomatic bacteriuria presenting with a prescription for an antibacterial from another health care practitioner.
  Interventions: Other: Advanced care

INTERVENTIONS:
Other: Advanced care — The pharmacist will assess for symptoms of urinary tract infection and, for patients in Arm 1, prescribe antibacterials when appropriate. For patients in Arm 2, pharmacists will ensure optimal therapy and adapt or perform therapeutic substitution when appropriate (or work with the patient to discontinue therapy or just put the prescription on file in instances where the patient is assessed to have asymptomatic bacteriuria for which treatment is inappropriate).

SUMMARY:
Pharmacists in some Canadian jurisdictions have recently been granted the ability to prescribe for uncomplicated urinary tract infections (UTIs). Therefore, the purpose of this study is to assess the impact that community pharmacists can have on the management of UTIs.

Pharmacists will identify potential study participants (patients) when they either present with symptoms of a UTI (such as difficulty or painful urination, increased frequency or urgency of urination) without a prescription for an antibiotic from another health care provider, or when they present with a prescription for an antibiotic from another health care provider to treat a UTI. For patients who consent to participate in the study, the pharmacist will screen for eligibility and assess for appropriateness of treatment.

If the patient does not already have a prescription for an antibiotic from another health care provider, the pharmacist will prescribe this for them if they meet certain criteria. If they do already have a prescription from another health care provider, the pharmacist will assess the appropriateness of the prescription and work with the patient to potentially change it to make it more appropriate, if necessary. If the pharmacist identifies any complicating factors that require a physician's assessment, the patient will be referred to their physician. The enrolled patients will also have a 2-week follow-up to assess for resolution of symptoms, unintended effects, and adherence to the treatment regimen. All data will be collected in a web-based registry that will maintain the patient's confidentiality outside of the pharmacy (i.e. patient initials, date of birth, and study identification (ID) number will be the only patient identifiers collected by the researchers). A patient satisfaction survey will also be administered via email.

DETAILED DESCRIPTION:
UTIs produce symptoms that may be unpleasant and distressing for patients and have the potential to lead to complications. It is also commonly misdiagnosed and treated inappropriately, resulting in unnecessary antimicrobial exposure and increased potential for adverse effects (including secondary infections, such as Clostridium difficile), as well as the selection of resistant pathogens. The incidence of UTI in women is 12% annually, with 50% of women reporting to have had a UTI by 32 years of age. Recurrence of infection occurs in 25% of women within 6 months of the first UTI, and this rate increases when more than one prior UTI has been experienced. In the elderly, the prevalence of asymptomatic bacteriuria (ASB) increases, with up to 20% of women at the age of 75 or older affected and up to 50% of institutionalized, non-catheterized elderly women affected, a finding that often results in the overuse of antibiotics. With bacterial resistance on the rise and a limited pipeline of antibacterials with novel mechanisms of action, antimicrobial stewardship has become imperative to maintain the effectiveness of available antimicrobials. Pharmacists are accessible primary care professionals that are well-positioned to take on a larger role in the management of medical conditions, including UTIs, and have an important role to play in antimicrobial stewardship. Therefore, it would be of great value to quantify the real-world impact of pharmacists providing care to patients with UTI, and then disseminate this information to inform best practice and policy change.

Design: prospective web-based registry Setting: ~40 community pharmacies in New Brunswick, Canada Patients: Any adult patient presenting to a pharmacy with symptoms suggestive of urinary tract infection (UTI) and assessed to be uncomplicated; or those presenting with a prescription for antibiotics from another healthcare provider for a UTI that are assessed to be uncomplicated or asymptomatic bacteriuria.

Intervention: Pharmacists will assess symptoms and prescribe antibiotics or perform prescription adaptation or therapeutic substitution, as necessary. They will also discontinue antibiotics for asymptomatic bacteriuria in cases where treatment is unnecessary. Follow-up will occur at 2 weeks to assess for clinical cure, as well as adverse reactions, adherence to the treatment regimen, early recurrence of infection, and other outcomes. Additional follow-up will occur as needed, and will also be captured in the registry.

Outcomes: The primary outcome will be clinical cure at 2 weeks. Secondary outcomes will include medications used, number and nature of pharmacist interventions, follow-ups conducted, patient adherence to initial recommendations and follow up, adverse events, treatment failures (including reasons for; such as adherence, delay in accessing care, missed baseline complicating factors, presence of a resistant organism, and complications such as pyelonephritis), and patient satisfaction.

Quality assurance: Data will be collected via a secure web-based portal. Data quality will be monitored by EPICORE Centre, University of Alberta, and site audits will be performed periodically.

Analytical plan: Most outcomes will be descriptive in nature. Target sample size of 750 patients over 8 months; this is a bit more than necessary for the primary outcome, but the intention is to also have enough power for analyses of some of the secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting without a prescription for antibacterials from another health care practitioner with symptoms of urinary tract infection that is found to be uncomplicated. Or patients presenting with a prescription for an antibacterial from another health care practitioner that is found to either have uncomplicated urinary tract infection or asymptomatic bacteriuria.

Exclusion Criteria:

* Patients with complicated urinary tract infections or symptoms suggestive of pyelonephritis or systemic illness.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to community pharmacies in New Brunswick, Canada with uncomplicated urinary tract infections.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Number of patients achieving clinical cure | 2 weeks
  Number of patients achieving sustained, full resolution of UTI symptoms, as described by the patient. This will be extracted from the registry database.

SECONDARY OUTCOMES:
Antibacterials used | 2 weeks
  The name of antibacterials used to treat infection and the number of instances that each antibacterial was used. This will be extracted from the registry database.
Pharmacist interventions | 2 weeks
  Number of pharmacist interventions collectively and individually by the following types: antibacterial initiation, modification of antibacterial regimen, discontinuation of antibacterial regimen, and referral to physician. These will be extracted from the registry database.
Adherence | 2 weeks
  Patient adherence to initial recommendations and follow up. Pharmacists will ask and document if the patient took the antibacterial as prescribed, if they missed one or two doses, if they missed 50% or more doses, or if they didn't take at all. The number of patients reporting each of these will be extracted from the registry database.
Number of treatment failures | 2 weeks
  Number of patients experiencing either treatment failure or recurrence of symptoms
Reasons for treatment failures | 2 weeks
  The likely contributory factors of the patients experiencing treatment failures, such as less than ideal adherence, missed baseline complicating factor, resistant pathogen, complication (such as pyelonephritis), delay in accessing care, other, or no identifiable reason. The number of times that each of these were considered potentially contributory to treatment failure will be extracted from the registry database.
Patient satisfaction as determined by the modified consultation satisfaction questionnaire | 2 weeks
  Satisfaction of patients with the service provided by the pharmacists as determined by patients' responses to survey questions on a likert scale.
Access to care | 2 weeks
  Time to seen by a pharmacist (Arm 1) or physician (Arm 2)
Adverse events | 2 weeks
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ross T Tsuyuki, BSc(Pharm), PharmD, MSc, Principal Investigator — Department of Medicine, University of Alberta; Daniel J Smyth, MD, Principal Investigator — Division of Infectious Diseases, Horizon Health Network
Locations (1):
- EPICORE Centre, University of Alberta, Edmonton, Alberta, Canada